CLINICAL TRIAL: NCT03603496
Title: Comparative Effectiveness of Post-Discharge Strategies for Hospitalized Smokers
Brief Title: Post-Discharge Smoking Cessation Strategies: Helping HAND 4
Acronym: HH4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000774/PHS
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Smoking Cessation
Keywords: Tobacco; Cessation; Hospitalization; eReferral; Interactive Voice Response; Tobacco Quitline
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Transitional Tobacco Care Management (TTCM) (Experimental): TTCM will provide 8 weeks of nicotine replacement therapy at hospital discharge and proactive contacts over 3 months delivered by automated IVR call. At each contact the patient is offered a return call from the hospital-based tobacco coach for counseling, medication advice, and coordination of care with the patient's outpatient health care team.
  Interventions: Behavioral: Transitional Tobacco Care Management (TTCM); Drug: Nicotine replacement therapy
- eReferral to State Tobacco Quitline (QL) (Active Comparator): Referral from hospital to the state Quitline will be made by the research team on behalf of each enrolled patient. Quitline staff will contact patient to offer up to 5 proactive telephone calls from a tobacco coach. Patient may also be eligible for NRT sample. Feedback from the quitline will be sent back to the patient's medical chart.
  Interventions: Behavioral: eReferral to State Tobacco Quitline (QL); Drug: Nicotine replacement therapy

INTERVENTIONS:
Behavioral: Transitional Tobacco Care Management (TTCM) — PTCM will provide sustained care after discharge by offering (1) 8 weeks of nicotine replacement therapy at no cost provided at hospital discharge and (2) up to 7 proactive contacts over 3 months delivered by automated IVR call, supplemented by text messaging and email (patient choice). At each contact the patient is offered a return call from the hospital-based tobacco coach who offer counseling, medication advice, and coordination of care with the patient's outpatient health care team.
  Arms: Transitional Tobacco Care Management (TTCM)
Behavioral: eReferral to State Tobacco Quitline (QL) — Referral from hospital to the state Quitline will be made by the research team on behalf of each enrolled patient. Feedback from the Quitline will be included in the patient's medical chart.
  Arms: eReferral to State Tobacco Quitline (QL)
Drug: Nicotine replacement therapy — Up to 8 weeks of nicotine replacement therapy provided at no cost to the patient.

SUMMARY:
This randomized controlled trial will compare the effectiveness of two models of post-discharge tobacco cessation treatment for adult smokers admitted to 3 U.S. hospitals.

DETAILED DESCRIPTION:
This multi-site randomized controlled trial (RCT) will compare the effectiveness of two models of post-discharge tobacco cessation treatment for adult smokers who are admitted to 3 large hospital systems in 3 U.S. regions (MA, PA, TN). All patients will receive guideline-based tobacco cessation treatment delivered in hospital by each site's existing Tobacco Treatment Service that is directed by a study investigator. Patients who plan to quit smoking after hospital discharge will be randomly assigned to 1 of 2 post-discharge tobacco treatment interventions and followed at 1, 3, and 6 months. One arm uses bidirectional electronic referral (eReferral) to the state tobacco quitline. The other arm, Personalized Tobacco Care Management (PTCM), combines proactive messages delivered by automated interactive voice response (IVR) phone calls, text messaging, and/or email with health coaching provided by a hospital-based tobacco counselor. Both groups will receive at least 1 month of nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current cigarette smoker (>=1 cigarette in the week before admission and >=1 cigarette/day when smoking at a baseline rate in the month prior to admission)
* Admitted to a study hospital
* Seen by hospital smoking counselor during inpatient stay
* Plans to try to quit smoking after hospital discharge

Exclusion Criteria:

* Inability to give informed consent or participate in counseling due to serious cognitive or psychiatric disorder (e.g., dementia, psychosis)
* Life expectancy <12 months
* Medical instability
* No reliable telephone access or inability to use telephone
* Non-English speaking
* Pregnant, breastfeeding, to planning to become pregnant in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1416 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital; Hilary A Tindle, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SS, Chang Y, Rigotti NA, Singer DE, Levy DE, Tyndale RF, Davis EM, Freiberg MS, King S, Wells QS, Tindle HA. Can Treatment Support Mitigate Nicotine Metabolism-Based Disparities in Smoking Abstinence? Secondary Analysis of the Helping HAND 4 Trial. Nicotine Tob Res. 2023 Aug 19;25(9):1575-1584. doi: 10.1093/ntr/ntad079. PMID 37209421
- [Derived] Rigotti NA, Chang Y, Davis EM, Regan S, Levy DE, Ylioja T, Kelley JHK, Notier AE, Gilliam K, Douaihy AB, Singer DE, Tindle HA. Comparative Effectiveness of Postdischarge Smoking Cessation Interventions for Hospital Patients: The Helping HAND 4 Randomized Clinical Trial. JAMA Intern Med. 2022 Aug 1;182(8):814-824. doi: 10.1001/jamainternmed.2022.2300. PMID 35759282
- [Derived] Rigotti NA, Schnitzer K, Davis EM, Regan S, Chang Y, Kelley JHK, Notier AE, Gilliam K, Douaihy A, Levy DE, Singer DE, Tindle HA. Comparative effectiveness of post-discharge strategies for hospitalized smokers: Study protocol for the Helping HAND 4 randomized controlled trial. Trials. 2020 Apr 16;21(1):336. doi: 10.1186/s13063-020-04257-7. PMID 32299470

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 708 patients were randomized to TTCM arm. 2 patients were excluded post-randomization but before hospital discharge and the start of the intervention and follow-up assessment due to not meeting eligibility criteria.
  708 patients were randomized to QL arm. 5 patients were excluded post-randomization but before hospital discharge and the start of the intervention and follow-up assessment due to not meeting eligibility criteria.
Groups:
- Transitional Tobacco Care Management (TTCM): TTCM will provide 8 weeks of nicotine replacement therapy at hospital discharge and proactive contacts over 3 months delivered by automated IVR call. At each contact the patient is offered a return call from the hospital-based tobacco coach for counseling, medication advice, and coordination of care with the patient's outpatient health care team.
  Transitional Tobacco Care Management (TTCM): TTCM will provide sustained care after discharge by offering (1) 8 weeks of nicotine replacement therapy at no cost provided at hospital discharge and (2) up to 7 proactive contacts over 3 months delivered by automated IVR call, supplemented by text messaging and email (patient choice). At each contact the patient is offered a return call from the hospital-based tobacco coach who offer counseling, medication advice, and coordination of care with the patient's outpatient health care team.
  Nicotine replacement therapy: Up to 8 weeks of nicotine replacement therapy provided at no cost to the patient.
Period: Overall Study
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Started | 706 | 703
Completed | 520 | 518
Not Completed | 186 | 185
Not completed — Death | 19 | 24
Not completed — Lost to Follow-up | 141 | 141
Not completed — Withdrawal by Subject | 26 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL) | Total
Number analyzed (Participants) | 706 | 703 | 1409
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 52 (12) | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391 | 393 | 784
  Male | 315 | 310 | 625
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 539 | 550 | 1089
  Black non-Hispanic | 116 | 100 | 216
  Hispanic | 39 | 43 | 82
  Asian/Pacific Islander | 4 | 3 | 7
  Other/unknown | 8 | 7 | 15
Cigarettes smoked per day, past 30 days [Mean (Standard Deviation); unit: cigarettes/day] | 16 (10) | 17 (11) | 16 (11)
Smoke 1st cigarette within 30 min of waking [Count of Participants; unit: Participants] — Measure of nicotine dependence. Smoking within 30 minutes of waking is associated with higher nicotine dependence.
  Participants | 547 | 563 | 1110

OUTCOME MEASURES:

1. Primary Outcome: Tobacco Abstinence, Biochemically Confirmed
Description: Participant self-report of no use of any tobacco product (cigarettes, cigars, little cigars, pipes, smokeless tobacco product) in the past 7 days AND either a saliva sample with a cotinine concentration <=10 ng/ml OR breath sample with a carbon monoxide concentration <=9 ppm.
Time Frame: 6 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 110 | 96
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); Two-stage multiple imputation techniques were used to estimate the missing smoking outcomes. 1st stage: we imputed missing data from surveys. 2nd stage: we imputed missing data from biochemical sample collection. Null hypothesis was no difference between arms in biochemically-validated past 7-day abstinence from cigarettes and other conventional tobacco products at 6-months. Sample of 1350 (675/group) was planned to detect a 6.5% difference (23.0% vs. 16.5%) with 84% power and 2-sided p<0.05; Test type: Superiority; p = .19, Chi-squared; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.92 to 1.50] — Comparing TTCM as numerator, QL as denominator (reference group)

2. Secondary Outcome: Tobacco Abstinence, Self-report
Description: Participant self-report of abstinence for the past 7 days from any tobacco product use (cigarettes, cigars, little cigars, pipes, smokeless tobacco product).
Time Frame: 1 month after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 291 | 246
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); Multiple imputation techniques were used to estimate the missing smoking outcomes. The null hypothesis was no difference between study arms; Test type: Superiority; p = .002, Chi-squared; Risk Ratio (RR) = 1.22, 95% CI 2-sided [1.08 to 1.35] — Numerator is TTCM, denominator (reference group) is QL

3. Secondary Outcome: Tobacco Abstinence, Self-report
Description: as for outcome 2
Time Frame: 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 276 | 218
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .001, Chi-squared; Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.09 to 1.37] — Numerator is TTCM, denominator (reference group) is QL

4. Secondary Outcome: Tobacco Abstinence, Self-report
Description: as for outcome 2
Time Frame: 6 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 234 | 202
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .079, Chi-squared; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.98 to 1.29] — Numerator is TTCM, denominator (reference group) is QL

5. Secondary Outcome: Engagement in Cessation Treatment
Description: Number of participants who report currently using tobacco treatment (defined as cessation medication or cessation counseling) at the 1 month post-discharge assessment.
Time Frame: 1 month after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 489 | 369
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); Participants lost to follow-up or with missing data are counted as having received no treatment. The null hypothesis was no difference between study arms; Test type: Superiority; p < .0001, Chi-squared; Risk Ratio (RR) = 1.32, 95% CI 2-sided [1.21 to 1.44]

6. Secondary Outcome: Engagement in Cessation Treatment
Description: Number of participants who report currently using tobacco treatment (defined as cessation medication or cessation counseling) at 3 month post-discharge assessment
Time Frame: 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 434 | 319
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < .0001, Chi-squared; Risk Ratio (RR) = 1.35, 95% CI 2-sided [1.23 to 1.50]

7. Secondary Outcome: Self-reported Continuous Tobacco Abstinence Since Hospital Discharge
Description: Number of participants who self-report having smoked no cigarettes and used no other tobacco products (cigars, little cigars, pipes, smokeless tobacco) since index hospital discharge
Time Frame: 6 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
Number analyzed (Participants) | 706 | 703
Participants | 120 | 91
Statistical Analysis 1: Comparison: Transitional Tobacco Care Management (TTCM) vs eReferral to State Tobacco Quitline (QL); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .033, Chi-squared; Risk Ratio (RR) = 1.31, 95% CI 2-sided [1.02 to 1.66] — Numerator is TTCM, denominator (reference group) is QL

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious adverse events and other (not including serious) adverse events were not monitored or systematically assessed in this trial. However, when attempting to conduct follow-up assessments, study staff learned of some deaths of study participants, usually from a family member or the electronic health record. We are able to report the number of deaths of participants that we learned about during the routine follow-up procedures.
Arm/Group | Transitional Tobacco Care Management (TTCM) | eReferral to State Tobacco Quitline (QL)
All-Cause Mortality (participants affected / at risk) | 19/706 | 24/703
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03603496/Prot_SAP_002.pdf